CLINICAL TRIAL: NCT05435937
Title: Partnering for Change (P4C) in Sweden - an Intersectional Collaborative Intervention to Create an Inclusive Learning Environment and Increased Conditions for Learning for Pupils at Risk of Unhealth, Exclusion and Low Academic Achievements
Brief Title: Partnering for Change in Sweden - Intervention to Increase Pupils' Engagement and Participation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Linkoeping University (Other Government)
Collaborators: Uppsala University (Other); Örebro University, Sweden (Other); Stockholm University (Other)
Responsible Party: Principal Investigator, Helene Lidstrom, Senior lecturer, Linkoeping University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HMV-2022-00021
Record Dates: First submitted 2022-06-22; First posted 2022-06-28 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Child Health
Keywords: Disabled Children; Special educational needs; Partnering for change; Universal design for learning; Participation; Tiered intervention model; Inclusive learning environment
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Non randomized control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- P4C-Swe intervention (Experimental): Pupils in participating classes will receive the Partnering for change (P4C) intervention
  Interventions: Behavioral: Partnering for change (P4C-Swe)
- Treatment as usual (Active Comparator): Treatment as usual is provided by the Student health services that consists of a school doctor, school nurse, psychologist and counselor, and staff with special educational competence
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: Partnering for change (P4C-Swe) — P4C focuses on the collaboration and a intersectional partnership between teachers and occupational therapists/special educators to create physical, social and learning environments that facilitate successful participation for all pupils. The intervention tiered model provides interventions in a school context in levels; class, group, and individual level to students with participation restrictions.
  Dynamic Performance Analysis (DPA), which focuses on pupils' occupational performance, is used in P4C model to identify and analyze were and why pupils' occupational performance is breaking down in school-based occupations in the natural context, followed by collaboration and coaching between the occupational therapist and teacher in setting up goals, planning, implementing and monitoring intervention at the different intervention levels, to support participation.
  Arms: P4C-Swe intervention
Behavioral: Treatment as usual — Treatment as usual is provided by the Student health services that consists of a school doctor, school nurse, psychologist and counselor, and staff with special educational competence
  Arms: Treatment as usual

SUMMARY:
This project implements an innovative and intersectional collaborative intervention model that addresses challenges that exist for children with special educational needs, who risk school failure, exclusion and poor health. The aim is to evaluate how the intervention model Partnering for Change (P4C) can be used to provide school-based services for creating an inclusive learning environment, and its effects on students 'conditions for learning, such as students' engagement and participation in school activities.

The study has a non-randomized controlled intervention study design with pre-, post- and follow-up measurements.

DETAILED DESCRIPTION:
This project implements an innovative and intersectional intervention school-based service delivery model that addresses challenges that exist for children with special educational needs who risk school failure, exclusion and poor health because of a) the lack of accommodations and support that meet their needs in school, b) the lack of knowledge and systematic work methods to create inclusive learning environments, and c) the lack of evidence-based school interventions. Despite investments in support for children with special needs, there is a large proportion of children who do not achieve educational goals due to low engagement, attendance at school, disability or mental ill-health or poor socio-economic environments. Poor educational results may lead to inequality in society, such as exclusion from higher education and/or labour market later in life. To meet these challenges, the following study project focuses on creating inclusive learning environments by implementing the Canadian evidence and school-based service delivery model Partnering for Change (P4C) in Swedish schools. The aim of the study is to investigate the P4C´s effect on children's prerequisites for learning and children's experiences of inclusive learning environment. P4C is based on universal design for learning and facilitate earlier identification of pupils who need support, and through early intervention, with a tiered model at class, group, and individual level, increase the conditions of learning. By implementing P4C, children with or without diagnosis, will have access to accommodations that match their needs. The results of a feasibility study, with preliminary results, shows good feasibility and acceptance for P4C in Swedish schools. Participants in current study are 20 classes (400 pupils, ages 6-12 years) (intervention and control classes), class teachers, occupational therapists and special educator teachers in student health services. A non-randomized controlled intervention study design with before, after and follow up measurements will answer how effective P4C is for children.

ELIGIBILITY:
Inclusion Criteria for group of pupils are:

1. that the school's pupils health service has access to an occupational therapist and/or special education teacher,
2. preschool class or primary school class years 1-6,
3. that school staff feel that there are pupils in class in special educational needs and/or in need of a more accessible learning environment
4. that the school principal and class teacher agree to participate in the study. -

Exclusion Criteria: None

-

Ages: 5 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 400 (Estimated)
Dates: Start 2022-02-10 (Actual); Primary Completion 2024-01-10 (Estimated); Study Completion 2024-06-10 (Estimated)

PRIMARY OUTCOMES:
Change in the Engagement Versus Disaffection With Learning: Teacher Report (EEL) | Baseline, four months, eleven months
  Engagement Versus Disaffection with Learning: Teacher Report (EEL) is a measure of school engagement from the perspective of a child's teacher. The EEL consists of four subscales across 25 items, and the teacher is instructed to rate on a four-point Likert-type scale, from 1 (Happens almost never) to 4 (Happens very often) how close each item describes the pupil.

SECONDARY OUTCOMES:
Change in the Swedish Child Health Utility 9D (CHU9D) | Baseline, four months, eleven months
  The CHU9D measures HRQoL by nine-dimensions: worried, sad, pain, tiredness, annoyed, school work/homework, sleep, daily routines, and ability to join in activities. Recall time is today, and each dimension has five severity levels e.g. I do not feel worried today, I feel very little worried today, I feel a little worried today, I feel pretty worried today or I feel very worried today.
Change in How I Feel About My School (HIFAMS) | Baseline, four months, eleven months
  The HIFAMS addresses seven questions of perceived well-being in the educational setting, including satisfaction with teachers, peers, classrooms, playgrounds, the transition to school, work and school in general. The HIFAMS uses a three-point Likert scale, where emotions are used to convey the responses Glad= a smiling face, Neutral=a neutral face, or Sad= a Sad face. The questionnaire is suitable for children aged 4 to 12 years.
Change in occupational performance in school-based occupations | During the four months intervention period
  Change in occupational performance, measured during observations of school-based occasion in natural context. Measured with a rating scale (1-10) 1=no performance 10= excellent performance. Measured once before and after implemented interventions for each identified performance break-down
Change in attainment of school-based occupational performance goals | During the four months intervention period
  Rated as attained, partly attained or not attained. Measured once before and after implemented interventions for each identified performance break-down
Change in School attendance | Baseline to eleven months
  Statistics registration of pupils attendance in percent per week during the data collection period (eleven months).
Change in School setting interview (SSI) | During the four months intervention period
  The School Setting Interview (SSI) is used only at individual level to examine the student-environment fit in a school setting. The SSI includes 16 items concerning everyday school activities and the pupils perceived need of adjustments is documented in each item. Each item is scored using a four-step rating scale; 4=Perfect fit, 3=Good fit, 2=<partly fit, and 1= Unfit. Measured once before and after implemented interventions for each identified performance break-down
Change in the Protocol of number of pupils with special educational needs | Baseline, four months, eleven months
  A study protocol has been developed to collect data of number of pupils who have access to adjustments and or support and number of pupils in need of adjustments and or support in each class.

CONTACTS AND LOCATIONS:
Overall Officials: Helene Lidström, PhD, Principal Investigator — Linkoeping University
Locations (3):
- Sweden (3):
  - Falu kommun, Falun
  - Karlskrona kommun, Karlskrona
  - Kinda kommun, Kisa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Baric VB, Yngve M, Holmefur M, Feldman I, Wilder J, Johansen K, Klang N, Lidstrom H, Borgestig M. Partnering for change (P4C) in Sweden- a study protocol of a collaborative school-based service delivery model to create inclusive learning environments. BMC Public Health. 2023 Nov 10;23(1):2219. doi: 10.1186/s12889-023-17053-0. PMID 37950243